CLINICAL TRIAL: NCT06639893
Title: Crestal Bone Loss in Mandibular Telescopic Implant Retained Overdenture with Milled Titanium, Milled Poly-ether Ketone Ketones and 3D Printed Chrome Cobalt Secondary Copings
Brief Title: Crestal Bone Loss in Mandibular Telescopic Overdentures. Overdenture with Milled Titanium, Milled Poly-ether Ketone Ketones and 3D Printed Chrome Cobalt Secondary Copings.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Minia University (Other)
Responsible Party: Principal Investigator, Moustafa mohamed el maghraby, Assistant lecturer of prosthodontics, Minia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Randomized clinical trial; 613 (Other: Ethical committe, El minia University)
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Telescopic Overdentures; Dental Implants; Customized Abutments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Milled Titanium secondary copings (Active Comparator)
  Interventions: Procedure: Telescopic overdenture
- 3D printed chrom cobalt copings. (Experimental)
  Interventions: Procedure: Telescopic overdenture
- Milled Poly-ether Ketone Ketones copings. (Experimental)
  Interventions: Procedure: Telescopic overdenture

INTERVENTIONS:
Procedure: Telescopic overdenture — Telescopic overdenture with two dental implants in intraforaminal area for mandible.

SUMMARY:
The objective of this clinical trial is to evaluate crestal bone loss every three months at time of overdenture insertion, 3, 6, 9, 12 months from overdenture use. Also, to evaluate prosthesis satisfaction.

All participants will receive conventional complete dentures, followed by two intraforaminal implants. After healing time, fabrication of secondary copings in all cases according to randomized groups for final overdenture insertion.

ELIGIBILITY:
Inclusion Criteria:

1. Sufficient remaining bone in height, width and thickness in the interforaminal area to allow installation of at least 3.3 mm diameter and 8 mm length implants.
2. Adequate amount of interarch space of at least 12mm.
3. Age range from 55 to 75 years old age.

Exclusion Criteria:

1. Systemic and metabolic diseases that may affect osseointegration.
2. Patients receiving bisphosphonates therapy.
3. Patients under radiotherapy or chemotherapy.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Crestal bone loss. | one year
  The aim of this study was to evaluate crestal peri implant bone loss in mandibular telescopic implant retained overdenture with milled titanium, milled poly-ether ketone ketones and 3D printed chrome cobalt secondary copings. Crestal bone loss evaluated every three months using standardized digital periapical radiograph at time of overdenture insertion, 3, 6, 9, and after 12 months from overdenture use.

CONTACTS AND LOCATIONS:
Locations (1):
- EL Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided